CLINICAL TRIAL: NCT01561599
Title: Pilot Study of BB3 to Improve Renal Function in Patients With Signs and Symptoms of Significant Renal Injury After Kidney Transplantation From Donors After Cardiac Death
Brief Title: Study on Delayed Graft Function Using Paired Kidneys
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Angion Biomedica Corp (Industry)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 004-09; 2010-019243-19 (EudraCT Number); 2R44DK078455-02 (NIH)
Record Dates: First submitted 2012-03-21; First posted 2012-03-23 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: Delayed Graft Function
Keywords: hepatocyte growth factor mimetic; hepatocyte growth factor(HGF); Delayed Graft Function (DGF); Kidney transplantation
MeSH Terms: conditions — Delayed Graft Function; Deafness, Autosomal Recessive 39 | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Normal saline (Placebo Comparator): Placebo
  Interventions: Drug: Normal Saline
- BB3 (Active Comparator): Small molecule mimetic of hepatocyte growth factor/scatter factor
  Interventions: Drug: BB3

INTERVENTIONS:
Drug: BB3 — Daily intravenous administration of 2mg/kg for 4 days
  Arms: BB3
Drug: Normal Saline — Daily intravenous administration for four (4) days. The volume of normal saline will vary by estimated weight.
  Arms: Normal saline

SUMMARY:
The study is designed to evaluate the safety and efficacy of an intravenously administered drug in recipients of kidneys from cardiac death donors who are risk for developing delayed graft function.

DETAILED DESCRIPTION:
Renal transplantation is the most effective and cost-efficient form of renal replacement therapy for a burgeoning population that presents with end-stage renal disease. Although organ donation has become a national priority, the gap between the number of patients awaiting a kidney versus the number of available kidneys continues to widen exponentially. In many countries within the European Union, utilization of "donation after cardiac death" (DCD) kidneys is steadily increasing, expanding the donor pool by > 50%. Given the high incidence of cardiac deaths in the US, aggressive pursuit of the DCD kidney pool could potentially reduce waitlist periods to months, if not days. Risk for delayed graft function (DGF) with the attendant risks for increased recipient morbidity, chronic allograft nephropathy and increased medical costs has however tempered DCD kidney utilization in this country. Development of strategies that limit normothermic reperfusion injury, promote renal repair, reduce the incidence and/or duration of DGF and improve long-term outcome can greatly enhance acceptance and recruitment of DCD kidneys. The study is designed to evaluate the safety and efficacy of an intravenously administered drug in recipients of kidneys from DCD donors who are risk for developing DGF. This trial is unique in that it compares drug versus placebo outcome in kidney recipients from the same donor with direct evaluation of function (creatinine clearance) in the graft.

ELIGIBILITY:
Inclusion Criteria

1. Subjects must sign the informed consent document prior to performance of any study related procedure including the Screening procedure.
2. Males and females ≥ 18 years of age.
3. Had renal transplantation due to end stage disease requiring chronic dialysis.
4. Study drug can be administered within 6 to 36 hours after transplantation.
5. Received kidney from donor after cardiac death.
6. DCD kidney fulfills the clinical site's criteria for transplantation.
7. Creatinine clearance from the transplanted kidney over a 2-hour collection period is <10 mL/min, OR no urine output OR average urine output of < 50 cc/H over 8 or more consecutive hours,, OR normal urine output following transplantation that diminished to average of < 50 cc/H over 8 or more consecutive hours, OR Creatinine reduction ratio 24 hours after transplantation to pre-transplantation is < 30%.
8. Dry weight ≤ 100 kg.
9. Women of child bearing potential have a negative pregnancy test prior to transplantation.
10. Women of child bearing potential (including perimenopausal women who have had a menstrual period within 1 year) must agree to use 2 forms of effective birth control regimen (at least one-barrier method) during the 28-day study period. Men must agree to use condoms during the study period; a condom with spermicide is considered a single barrier.
11. In the opinion of the Investigator, the subject is capable of understanding and complying with the protocol.

Exclusion Criteria

1. Mean arterial pressure <40 mmHg or cardiac index <1.8 L/min/m2.
2. Recipient of multiple organ transplantation or scheduled for multiple organ transplantation.
3. Recipient of kidney from a pediatric donor age 10 years or less.
4. Recipient age > 75 years.
5. Patients with ASA 4 or 5
6. Patients with chronic obstructive pulmonary disease (COPD) GOLD IV
7. Has measurable donor-specific antibody or positive cross-match requiring deviation from standard immunosuppressive therapy.
8. Currently participating in or has participated in an investigational drug or medical device study within 30 days or five half-lives, whichever is longer, prior to enrolment into this study.
9. Concurrent sepsis or active bacterial infection.
10. Have an active malignancy or history of solid, metastatic or hematologic malignancy with the exception of basal or squamous cell carcinoma of the skin that has been removed.
11. Women of child bearing potential who is breast feeding.
12. History of positive HIV test.
13. History of rheumatoid arthritis.
14. History of proliferative retinopathy or laser surgery for retinopathy.
15. Subjects who have a penicillin allergy.
16. Subjects who require the cytochrome P450 1A2 (CYP1A2) inhibitors, or are receiving ciprofloxacin and fluvoxamine (Luvox®).
17. Subject is unwilling or unable to comply with the protocol or to cooperate fully with the Investigator or the site personnel.
18. Subject is not deemed medically stable for the study in the opinion of the Investigator or the subject's primary nephrologist.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-08; Primary Completion 2016-02 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
creatinine clearance | 7 days
  The primary analysis to assess the activity of BB3 compared to placebo will be the mean difference in creatinine clearance over time using selective 24-hour urine collections from the transplanted kidney from the first infusion of study drug through day 7 post-transplant.

SECONDARY OUTCOMES:
Urine production | 28 days
  Median time (days) until production of ≥1 litre urine over a 24-hour period, i.e. median number of days following the first infusion of study drug until the first day (08:00 - 08:00) that urine production was ≥1 litre over a 24-hour period.
Creatinine clearance | 28 days
  Calculated creatinine clearance at days 14 and 28
Incidence of delayed graft function | 7 days
  Incidence of delayed graft function (required dialysis due to inadequate renal function during the first 7 days after transplantation).
Number of dialysis sessions | 28 days
  Number of dialysis sessions through day 7, 14, and 28
Mean total daily urine output | 14 days
  Mean total daily urine output through day 14
Daily serum creatinine | 7 days
  Daily serum creatinine at days 1 to 7
Mean serum creatinine | 28 days
  Mean serum creatinine at days 4, 7, 10, 14, and 28
Length of hospitalization following transplantation | 28 days
  Length of hospitalization following transplantation
Follow-up on graft survival and function | 12 months
  Results of the 6- and 12-month follow-up on graft survival and function will be summarized as an addendum to the final clinical study report

CONTACTS AND LOCATIONS:
Locations (3):
- Maastricht University Medical Center, Minderbroedersberg, Maastricht, Netherlands
- Hospital Clínico San Carlos, San Carlos, Madrid, Spain
- The Newcastle Upon Tyne Hospital, Newcastle, Metropolitan County of Tyne and Wear, United Kingdom